CLINICAL TRIAL: NCT04441112
Title: Intraarticular Injections of the Hip and Knee With Triamcinolone Versus Ketorolac: A Randomized Controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Saint Alphonsus Regional Medical Center (Other)
Responsible Party: Principal Investigator, Kevin Jurgensmeier, Medical Student, Saint Alphonsus Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SaintAlphonsusRMC
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Arthritis Knee; Arthritis of Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ketorolac Intraarticular Hip Injection (Experimental): Patients will receive an intraarticular hip injection with ketorolac.
  Interventions: Drug: Ketorolac Intraarticular Injection
- Triamcinolone Intraarticular Hip Injection (Active Comparator): Patients will receive an intraarticular hip injection with triamcinolone.
  Interventions: Drug: Triamcinolone Intraarticular Injection
- Ketorolac Intraarticular Knee Injection (Experimental): Patients will receive an intraarticular knee injection with ketorolac.
  Interventions: Drug: Ketorolac Intraarticular Injection
- Triamcinolone Intraarticular Knee Injection (Active Comparator): Patients will receive an intraarticular knee injection with triamcinolone.
  Interventions: Drug: Triamcinolone Intraarticular Injection

INTERVENTIONS:
Drug: Ketorolac Intraarticular Injection — Injections will be given under ultrasound guidance with one of two possible medications.
  Arms: Ketorolac Intraarticular Hip Injection; Ketorolac Intraarticular Knee Injection
Drug: Triamcinolone Intraarticular Injection — Injections will be given under ultrasound guidance with one of two possible medications.
  Arms: Triamcinolone Intraarticular Hip Injection; Triamcinolone Intraarticular Knee Injection

SUMMARY:
Clinicians commonly utilize intraarticular injections to treat symptomatic primary arthritis. Steroid injections are common yet have immune-modulating effects and can alter gene expression which may delay definitive arthroplasty and further damage cartilage. Non-steroidal anti-inflammatory (NSAID) injections may offer a safer profile due to their differing mechanism of action; however, there is a relative dearth of information regarding their efficacy. This non-inferiority study compares the effectiveness of triamcinolone versus ketorolac in treating symptoms of moderate to advanced primary osteoarthritis of the hip and knee.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, radiographically proven degenerative joint disease in the hip or knee

Exclusion Criteria:

* recent injection in the hip or knee within the previous 3 months
* history of traumatic osteoarthritis or ligamentous reconstruction
* chronic narcotic use
* history of inflammatory or neuropathic arthropathy
* pregnant and/or nursing women
* allergy or strong reaction to study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale (Baseline to One Week Post-injection) | Comparing baseline to one week post-injection
  Pain Score
Change in Visual Analogue Scale (Baseline to One Month Post-injection) | Comparing baseline to one month post-injection
  Pain Score
Change in Visual Analogue Scale (Baseline to Three Months Post-injection) | Comparing baseline to three months post-injection
  Pain Score
Change in PROMIS Global Health Scores (Baseline to One Week Post-injection) | Comparing baseline to one week post-injection
  Overall patient wellbeing
Change in PROMIS Global Health Scores (Baseline to One Month Post-injection) | Comparing baseline to one month post-injection
  Overall patient wellbeing
Change in PROMIS Global Health Scores (Baseline to Three Months Post-injection) | Comparing baseline to three months post-injection
  Overall patient wellbeing
Change in Knee Injury and Osteoarthritis Outcome Score Jr. (Baseline to One Week Post-injection) | Comparing baseline to one week post-injection
  Functionality and pain of affected knee
Change in Knee Injury and Osteoarthritis Outcome Score Jr. (Baseline to One Month Post-injection) | Comparing baseline to one month post-injection
  Functionality and pain of affected knee
Change in Knee Injury and Osteoarthritis Outcome Score Jr. (Baseline to Three Months Post-injection) | Comparing baseline to three months post-injection
  Functionality and pain of affected knee
Change in Hip Injury and Osteoarthritis Outcome Score Jr. (Baseline to One Week Post-injection) | Comparing baseline to one week post-injection
  Functionality and pain of affected hip
Change in Hip Injury and Osteoarthritis Outcome Score Jr. (Baseline to One Month Post-injection) | Comparing baseline to one month post-injection
  Functionality and pain of affected hip
Change in Hip Injury and Osteoarthritis Outcome Score Jr. (Baseline to Three Months Post-injection) | Comparing baseline to three months post-injection
  Functionality and pain of affected hip

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Jurgensmeier, BS, Principal Investigator — Student Investigator at Saint Alphonsus Regional Medical Center; Steven B Daines, MD, Study Chair — Surgeon at Saint Alphonsus Regional Medical Center
Locations (1):
- Saint Alphonsus Regional Medical Center, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan currently decided.

REFERENCES:
- [Derived] Jurgensmeier K, Jurgensmeier D, Kunz DE, Fuerst PG, Warth LC, Daines SB. Intra-articular Injections of the Hip and Knee With Triamcinolone vs Ketorolac: A Randomized Controlled Trial. J Arthroplasty. 2021 Feb;36(2):416-422. doi: 10.1016/j.arth.2020.08.036. Epub 2020 Aug 22. PMID 32950343